CLINICAL TRIAL: NCT04981119
Title: An Observational Study Obtaining Solid Tumor Tissue From Participants and Apheresis for CAR T-Cell Therapy Manufacturing
Brief Title: Solid Tumor Analysis for HLA Loss of Heterozygosity (LOH) and Apheresis for CAR T- Cell Manufacturing
Acronym: BASECAMP-1
Status: Recruiting | Type: Observational
Sponsor: A2 Biotherapeutics Inc. (Industry)
Collaborators: Tempus AI (Industry)
Responsible Party: Sponsor
Other Study IDs: A2B101-101
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor, Adult; Colorectal Cancer; Non Small Cell Lung Cancer; Pancreatic Cancer; CRC; NSCLC; Pancreas Cancer; Mesothelioma; Ovarian Cancer; Ovarian Neoplasms; Ovarian Carcinoma; Mesothelioma, Malignant; Mesothelioma; Lung; Cancer; Triple Negative Breast Cancer (TNBC); Renal Cell Carcinoma (Kidney Cancer); Head and Neck Squamous Cell Carcinoma HNSCC
Keywords: CAR T Cell Therapy; Next Generation Sequencing; Leukapheresis; Apheresis; Immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Mesothelioma; Ovarian Neoplasms; Mesothelioma, Malignant; Neoplasms; Triple Negative Breast Neoplasms; Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Blood Component Removal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood or saliva, or buccal swabs will be obtained to determine germline HLA type as wells a germline comparison for tumor comparison. Archived tumor tissue samples will be obtained for NGS to determine LOH status of tumor tissue. DNA and RNA will be retained for enrolled participants only, if repeat testing if required. No further genetic testing will be performed on these samples.
  Peripheral Blood Mononuclear Cells (PBMCs) will be collected for enrolled subjects, enriched for T cells and cryopreserved for future manufacturing of an A2 Biotherapeutics, Inc. CAR T-cell therapy upon participant relapse. No further genetic testing will be performed on this sample.
  Archival tumor slides will be obtained for immunohistochemistry (IHC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Apheresis — Apheresis procedure performed for collection of PBMCs.
Diagnostic Test: Next Generation Sequencing (NGS) — NGS on tumor tissue and a matched normal sample for loss of heterozygosity in tumor tissue and tumor tissue markers.
Diagnostic Test: Long Range NGS HLA typing — Long range NGS on whole blood to determine germline HLA type.

SUMMARY:
Objective:

To collect information on how often a solid tumor cancer might lose the Human Leukocyte Antigen (HLA) by next generation sequencing and perform apheresis to collect and store an eligible participant's own T cells for future use to make CAR T-Cell therapy for their disease treatment.

Design:

This is a non-interventional, observational study to evaluate participants with solid tumors with a high risk of relapse for incurable disease. No interventional therapy will be administered on this study. Some of the information regarding the participant's tumor analysis may be beneficial to management of their disease. Participants that meet all criteria may be enrolled and leukapheresed (blood cells collected). The participant's cells will be processed and stored for potential manufacture of CAR T-cell therapy upon relapse of their cancer.

DETAILED DESCRIPTION:
Background:

Human Leukocyte Antigen (HLA) is a protein on the outside of cells that allows the immune system to recognize it's own cells as normal and leave them alone or respond if infected with a virus or bacteria, or a tumor cell. HLA might not be expressed normally on cancer cells. This may be why cancer can grow undetected by the immune system and is referred to as a tumor escape mechanism. Tumor escape can occur for many reasons, but one reason is Loss of Heterozygosity (LOH). LOH is the loss of one of the genes that encodes HLA protein. A2 Biotherapeutics, Inc. (A2 Bio) is developing therapies to recognize, target, and kill cancer cells that do not express HLA normally, and minimize any damage to normal cells that express normal HLA.

Once participants are identified as having LOH on their tumors, apheresis, a procedure to separate and collect white blood cells will be performed. It is the first required step in manufacturing CAR T-cell therapy. The collected T cells will be stored for patients that are likely to benefit from CAR T-cell therapy during their disease care.

Study Design:

Approximately 1000 participants will be screened for part 1 of the study, including HLA typing, approximately 500 participants will have NGS testing on their tumor samples and be followed for up to 2 years on the study, and up to 200 participants will be screened for part 2 of the study and enrolled if eligible and apheresed and be followed for up to 2 years on the study.

Participants will be screened (Part 1) for HLA type, and based on results, participants will have archived tumor tissue tested by next generation sequencing (NGS) and be followed for up to 2 years. Based on the tumor NGS results, participants will be apheresed (Part 2) for Peripheral Blood Mononuclear Cell (PBMC) collection to store their T cells for a future interventional study upon relapse.

Each participant will proceed through the following study periods:

* Screening (Part 1 and 2)
* Enrollment (Apheresis)
* Post Apheresis safety follow-up (Day 7)
* Two-year long term follow-up

ELIGIBILITY:
Key Eligibility Criteria (additional criteria may apply) Part 1 Key Inclusion Criteria

1. Pathologically confirmed solid tumors, e.g., Colorectal Cancer (CRC), Non-Small Cell Lung Cancer (NSCLC), or Pancreatic Cancer (PANC), that is metastatic, unresectable locally advanced, or in the Investigator's opinion the subject is high risk for incurable relapse within two years.

Part 1: Key Exclusion Criteria

1. History of any of other malignancy in the past 5 years other than non-melanoma skin carcinoma, low grade localized prostate cancer, superficial bladder cancer, ductal carcinoma in situ (CIS) of the breast, CIS of the Cervix, or Stage I uterine cancer.
2. Prior allogeneic stem cell transplant.
3. Prior solid organ transplant.

Part 2 : Key Inclusion Criteria

1. Pathologically confirmed solid tumors, e.g., Colorectal Cancer (CRC), Non-Small Cell Lung Cancer (NSCLC), Pancreatic Cancer (PANC), Mesothelioma, or Ovarian Cancer (OVAC) that is metastatic, unresectable locally advanced, or in the Investigator's opinion the subject is high risk for incurable relapse within two years.
2. Participants are germline HLA-A*02 heterozygous confirmed by HLA typing.
3. Primary tumor tissue showing LOH of HLA-A*02 by NGS testing.
4. Eastern Cooperative Oncology Group (ECOG) 0 or 1 performance status.

Part 2: Key Exclusion Criteria

1. History of any of other malignancy in the past 5 years other than non-melanoma skin carcinoma, low grade localized prostate cancer, superficial bladder cancer, ductal carcinoma in situ (CIS) of the breast, CIS of the Cervix, or Stage I uterine cancer.
2. Prior allogeneic stem cell transplant.
3. Prior solid organ transplant.
4. Participants who have received any cancer therapy on any investigational therapy for any indication, including but not limited to chemotherapy, small molecules, monoclonal antibodies, or radiotherapy (with bone marrow impact) within 2 weeks of planned apheresis or 3 half-lives, whichever is shorter.
5. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment necessitating specific treatment, or any major episode of infection requiring treatment with Intravenous (IV) antimicrobials (e.g., IV antibiotics) or hospitalization (relating to completion of antibiotic course).
6. Has known active central nervous system metastases. Subjects with previously treated brain metastases may participate upon medical monitor agreement.
7. In the Investigator's judgement, any other condition or reason the subject would not complete the required study visits and procedures, and follow up visits, or comply with the study requirements for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Colorectal Cancer (CRC), Non-Small Cell Lung Cancer (NSCLC), Pancreatic Cancer (PANC), mesothelioma, or Ovarian Cancer (OVAC) that is metastatic, unresectable locally advanced, or in the Investigator's opinion the subject is high risk for incurable relapse within two years, germline HLA-A*02 heterozygous, and have confirmed somatic LOH.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-29 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who can enroll in an A2 Biotherapeutics, Inc. CAR T-cell therapy study after undergoing apheresis | up to 2 years
  Participants will be followed for their status of enrollment on an A2 Biotherapeutics, Inc. interventional study
Percentage of screened participants experiencing loss of heterozygosity (LOH) of HLA-A*02 identified by next generation sequencing | Screening
  Percentage of participants experiencing LOH will be calculated based on NGS results

SECONDARY OUTCOMES:
Percentage of enrolled participants who experience an adverse event (AE) related to apheresis | 7 days
  Adverse events will be collected and monitored for relatedness to apheresis during the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Eric W Ng, MD, FAAP, Study Director — A2 Biotherapeutics Inc.
Locations (16):
- United States (16):
  - Banner Health, Gilbert, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - City of Hope, Duarte, California
  - University of California San Diego, La Jolla, California
  - Stanford University, Palo Alto, California
  - UCLA Medical Center, Santa Monica, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital/Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - NYU Langone Medical Center, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Viale PH. The American Cancer Society's Facts & Figures: 2020 Edition. J Adv Pract Oncol. 2020 Mar;11(2):135-136. doi: 10.6004/jadpro.2020.11.2.1. Epub 2020 Mar 1. No abstract available. PMID 33532112
- [Background] Hamburger AE, DiAndreth B, Cui J, Daris ME, Munguia ML, Deshmukh K, Mock JY, Asuelime GE, Lim ED, Kreke MR, Tokatlian T, Kamb A. Engineered T cells directed at tumors with defined allelic loss. Mol Immunol. 2020 Dec;128:298-310. doi: 10.1016/j.molimm.2020.09.012. Epub 2020 Oct 1. PMID 33012527
- [Background] Hwang MS, Mog BJ, Douglass J, Pearlman AH, Hsiue EH, Paul S, DiNapoli SR, Konig MF, Pardoll DM, Gabelli SB, Bettegowda C, Papadopoulos N, Vogelstein B, Zhou S, Kinzler KW. Targeting loss of heterozygosity for cancer-specific immunotherapy. Proc Natl Acad Sci U S A. 2021 Mar 23;118(12):e2022410118. doi: 10.1073/pnas.2022410118. PMID 33731480
- [Background] Perera J, Mapes B, Lau D, et al. Detection of human leukocyte antigen class I loss of heterozygosity in solid tumor types by next-generation DNA sequencing. J Immunother Cancer. 2019, 7(Suppl 1):P103
- [Background] Beroukhim R, Mermel CH, Porter D, Wei G, Raychaudhuri S, Donovan J, Barretina J, Boehm JS, Dobson J, Urashima M, Mc Henry KT, Pinchback RM, Ligon AH, Cho YJ, Haery L, Greulich H, Reich M, Winckler W, Lawrence MS, Weir BA, Tanaka KE, Chiang DY, Bass AJ, Loo A, Hoffman C, Prensner J, Liefeld T, Gao Q, Yecies D, Signoretti S, Maher E, Kaye FJ, Sasaki H, Tepper JE, Fletcher JA, Tabernero J, Baselga J, Tsao MS, Demichelis F, Rubin MA, Janne PA, Daly MJ, Nucera C, Levine RL, Ebert BL, Gabriel S, Rustgi AK, Antonescu CR, Ladanyi M, Letai A, Garraway LA, Loda M, Beer DG, True LD, Okamoto A, Pomeroy SL, Singer S, Golub TR, Lander ES, Getz G, Sellers WR, Meyerson M. The landscape of somatic copy-number alteration across human cancers. Nature. 2010 Feb 18;463(7283):899-905. doi: 10.1038/nature08822. PMID 20164920
- [Background] McGranahan N, Rosenthal R, Hiley CT, Rowan AJ, Watkins TBK, Wilson GA, Birkbak NJ, Veeriah S, Van Loo P, Herrero J, Swanton C; TRACERx Consortium. Allele-Specific HLA Loss and Immune Escape in Lung Cancer Evolution. Cell. 2017 Nov 30;171(6):1259-1271.e11. doi: 10.1016/j.cell.2017.10.001. Epub 2017 Oct 26. PMID 29107330
- [Background] Priestley P, Baber J, Lolkema MP, Steeghs N, de Bruijn E, Shale C, Duyvesteyn K, Haidari S, van Hoeck A, Onstenk W, Roepman P, Voda M, Bloemendal HJ, Tjan-Heijnen VCG, van Herpen CML, Labots M, Witteveen PO, Smit EF, Sleijfer S, Voest EE, Cuppen E. Pan-cancer whole-genome analyses of metastatic solid tumours. Nature. 2019 Nov;575(7781):210-216. doi: 10.1038/s41586-019-1689-y. Epub 2019 Oct 23. PMID 31645765
- See also: A2 Bio website — http://www.a2bio.com